CLINICAL TRIAL: NCT01166256
Title: Prospective, Open-labeled, Randomized Controlled Trial of Comparison Between High-flow Nasal Cannula System and Non-invasive Ventilation in Acute Hypoxemic Respiratory Failure
Brief Title: Comparison Between High-flow Nasal Cannula System and Non-invasive Ventilation in Acute Hypoxemic Respiratory Failure
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Chae-Man Lim, Department of Pulmonary and Critical Care Medicine, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFNCinAHRF
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

ARMS (2):
- High-flow nasal cannula (Experimental): In this arm,patients with acute hypoxemic respiratory failure were treated with high-flow nasal cannula system(Optiflow, Fisher & Paykel, Auckland, New Zealand) to achieve SpO2 >92% or PaO2 >65 mmHg.
  Interventions: Device: High flow nasal cannula system
- Non-invasive ventilation (Active Comparator): In this arm, patients with acute hypoxemic respiratory failure is treated with the bi-level positive airways pressure mode (BiPAP Vision, Respironics Inc., Murrysville, PA) S/T mode to achieve SpO2 >92% or PaO2 >65 mmHg.
  Interventions: Device: Non-invasive ventilation

INTERVENTIONS:
Device: Non-invasive ventilation — Noninvasive ventilation: The inspiratory(IPAP) and expiratory positive airways pressure (EPAP), and the levels of FiO2 is set achieve SpO2 >92% or PaO2 >65 mmHg.
  Other Names: (BiPAP Vision, Respironics Inc., Murrysville, PA)
  Arms: Non-invasive ventilation
Device: High flow nasal cannula system — High flow nasal cannula system: FiO2 and flow rate of oxygen is set to achieve SpO2 >92% or PaO2 >65 mmHg.
  Other Names: Optiflow(Fisher & Paykel, Auckland, New Zealand)
  Arms: High-flow nasal cannula

SUMMARY:
Acute hypoxemic respiratory failure may require invasive mechanical ventilation. However, invasive mechanical ventilation is associated with a variety of complications. Non-invasive ventilation has been presented as an alternative treatment but controversy remains. The investigators hypothesize that high-flow nasal cannula system is effective enough to prevent intubation in acute hypoxemic respiratory failure and not inferior to non-invasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* patients with acute hypoxemic respiratory failure

Exclusion Criteria:

* age < 18 years
* hypercapnia (arterial carbon dioxide tension (PaCO2) >45mmHg) at admission
* need for emergency intubation, including cardiopulmonary resuscitation
* recent esophageal, facial or cranial trauma or surgery
* severely decreased consciousness (Glasgow coma score <11)
* cardiogenic shock or severe hemodynamic instability
* systolic blood pressure <90 mmHg associated with decreased urinary output(<20 mL.h-1) despite fluid repletion and use of vasoactive agents
* lack of co-operation
* altered mental status with decreased consciousness and/or evidence of inability to understand or lack of willingness to co-operate with the procedures
* tracheotomy or other upper airway disorders
* severe ventricular arrhythmia or active myocardial ischemia
* active upper gastrointestinal bleeding
* inability to clear respiratory secretions
* more than one severe organ dysfunction in addition to respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Success rate of treatment in two groups | up to 28 days
  Successful treatment is to avoid intubation and achieve PaO2 >75 mmHg without respiratory distress for 24 hours while spontaneously breathing oxygen provided by a Venturi device at FiO2 0.50.

SECONDARY OUTCOMES:
compliance of treatment | up to 28 days
  Withdrawl of non-invasive ventilation or high-flow nasal cannula system without intubation because of intolerance
adverse event | up to 28 days
hospital length of stay | up to 90 days
Hospital mortality | up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Chae-Man Lim, M.D., Study Chair — Department of Pulmonary and Critical Care Medicine, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea